CLINICAL TRIAL: NCT06253858
Title: Ultrasound (US) Guided External Ventricular Catheter Placement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Chris Zacko, Chris Zacko, MD Professor and Vice Chair for Quality, Department of Neurosurgery, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00022095
Record Dates: First submitted 2024-01-22; First posted 2024-02-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-04

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Catheter placement with Solopass system (Experimental): The Solopass US system will be used during catheter placement procedure to guide the placement of the catheter.
  Interventions: Device: Catheter Placement with Solopass System

INTERVENTIONS:
Device: Catheter Placement with Solopass System — This device is used as a guidance for placing a brain catheter to target the brain ventricles and decrease multiple brain passes, incorrect deployment and malfunctioning of the drain.

SUMMARY:
To assess the accuracy the SOLOPASS® System US based in the placement of external ventricular drain into the cranial cavity. This study will aim at evaluating the proposed efficacy of the device in targeting the brain ventricles and decrease multiple brain passes, incorrect deployment and malfunctioning of the drain.

ELIGIBILITY:
Inclusion Criteria:

* Decision made to perform the procedure by the primary consultant
* Age 18 or older
* Neuro ICU stay
* Newly diagnosed hydrocephalus
* Has a recent CT within the past 24 hrs
* Normal platelets and coagulation profile
* No active infection or currently on antibiotics
* The targeted fluid compartment has more than 50 percent CSF vs blood by CT scan imaging

Exclusion Criteria:

* Age <18
* Not in Neuro ICU setting
* Previous placement of a ventricular catheter
* More than 50 percent of the fluid compartment is filled with blood by CT scan
* Time to include in the trial prohibited by clinical personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Average number of passes needed to place the catheter in each subject. | 0 minutes
  Measured by the number of passes needed to place the catheter. If the first attempt fails, another US sweep will be performed, and another attempt will be performed. If that fails, then the procedure will be aborted.

SECONDARY OUTCOMES:
Post procedure imaging accuracy of the placement of the EVD will be performed by reviewing post procedure imaging using the Kakarla scoring system | up to 7 days
  Grade 1 means optimal placement in the ipsilateral frontal horn or third ventricle; Grade 2 means a functional placement in the contralateral lateral ventricle or no eloquent cortex; and Grade 3 means suboptimal placement in the eloquent cortex or nontarget cerebrospinal fluid space, with or without functional drainage

OTHER OUTCOMES:
Length of time of the procedure | Up to three hours
  Number of minutes necessary to complete the procedure placement of the catheter
Number of revision | up to 7 days
  Quantity of revisions due to the catheter malfunction
Number of subjects with Cerebrospinal fluid (CSF) infection | up to 7 days
  CSF will be collected as part of standard of care after the procedure and tested for infection.
Number of subjects with Superficial surgical site infection (SSI) | up to 7 days
  (The CDC defines SSI as deep and superficial. A superficial incisional SSI is an infection in the area of the skin where the incision was made. A deep incisional SSI occurs beneath the incision area in the muscle and the tissues surrounding the muscles. Signs to be monitored daily and put in a checklist will include redness, pain, unexplained fever source, pain, warmth, pus or swelling.)
Longevity of the device function | up to 7 days
  Number of days until a subsequent catheter is placed

CONTACTS AND LOCATIONS:
Overall Officials: J C Zacko, MD, Principal Investigator — Milton S. Hershey Medical Center